CLINICAL TRIAL: NCT06319027
Title: Phase II Glioblastoma Accelerated Biomarkers Learning Environment Trial (GABLE)
Brief Title: Identifying Findings on Brain Scans That Could Help Make Better Predictions About Brain Cancer Progression, The GABLE Trial
Acronym: GABLE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EAF223; NCI-2023-08557 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAF223 (Other: ECOG-ACRIN Cancer Research Group); EAF223 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma, IDH-Wildtype
MeSH Terms: conditions — Glioblastoma | interventions — fluciclovine F-18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (DSC-MRI, fluciclovine F18 PET, MR spectroscopy) (Experimental): Patients receive a gadolinium-based contrast agent and undergo DSC-MRI scans at 4 and 8 weeks after completion of SOC radiation therapy. Patients with evidence of disease progression then undergo MR spectroscopy or receive fluciclovine F18 IV and undergo PET scan within 12 weeks of SOC radiation therapy completion.
  Interventions: Procedure: Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging; Other: Fluciclovine F18; Drug: Gadolinium-Chelate; Procedure: Magnetic Resonance Spectroscopy; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging — Undergo DSC-MRI
  Other Names: DSC; DSC-MRI; Dynamic Susceptibility Contrast-Enhanced MRI; DYNAMIC SUSCEPTIBILITY-CONTRAST MRI
Other: Fluciclovine F18 — Given IV
  Other Names: (18F)Fluciclovine; (18F)GE-148; 18F-Fluciclovine; [18F]FACBC; Anti-(18f)FABC; Anti-1-Amino-3-[18F]Fluorocyclobutane-1-Carboxylic Acid; Anti-[18F] FACBC; Axumin; Fluciclovine (18F); FLUCICLOVINE F-18; GE-148 (18F); GE-148 F-18
Drug: Gadolinium-Chelate — Receive gadolinium-based contrast agent
  Other Names: Gadolinium Coordination Complex; Gadolinium-based Contrast Agent; Gadolinium-Chelant Complex
Procedure: Magnetic Resonance Spectroscopy — Undergo MR spectroscopy
  Other Names: NMR Spectroscopy; NUCLEAR MAGNETIC RESONANCE SPECTROSCOPY; Spectroscopy, MR; Spectroscopy, NMR; Spectroscopy, Nuclear Magnetic Resonance
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase II trial studies whether different imaging techniques can provide additional and more accurate information than the usual approach for assessing the activity of tumors in patients with newly diagnosed glioblastoma. The usual approach for this currently is magnetic resonance imaging (MRI). This study is trying to learn more about the meaning of changes in MRI scans after treatment, as while the appearance of some of these changes may reflect progressing tumor, some may be due the treatment. Dynamic susceptibility contrast (DSC)-MRIs, along with positron emission tomography (PET) and/or magnetic resonance (MR) spectroscopy, may help doctors tell which changes are a reflection of the treatment and which changes may be due to progressing tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. For each biomarker (dynamic susceptibility contrast-enhanced MR Imaging, fluciclovine F18 [18F-fluciclovine] PET, MR spectroscopy), to evaluate whether the biomarker can stratify patients with newly diagnosed glioblastoma (GBM) that have progressive enhancement within 12 weeks post-radiation therapy (XRT) into risk groups based on overall survival.

SECONDARY OBJECTIVES:

I. To evaluate whether each biomarker (dynamic susceptibility contrast-enhanced MR Imaging, 18F-fluciclovine PET, MR spectroscopy) can predict final determination of pseudo-progression (PsP) versus (vs.) true progression on follow-up MR imaging as evaluated by a semi-automated central reading process and by institutional radiologist readings.

II. To evaluate whether a prediction model that incorporates multiple biomarkers can discriminate patients with progressive enhancement within 12 weeks post-XRT into high and low risk groups for overall survival.

III. To evaluate whether clinical and imaging biomarkers are predictive of overall and progression-free survival in patients who do not show progressive enhancement within 12 weeks post-XRT.

EXPLORATORY OBJECTIVE:

I. To determine how different methods of defining PsP vs. true progression on imaging relate to patient survival.

OUTLINE:

Patients receive a gadolinium-based contrast agent and undergo DSC-MRI scans at 4 and 8 weeks after completion of standard of care (SOC) radiation therapy. Patients with evidence of disease progression then undergo MR spectroscopy or receive fluciclovine F18 intravenously (IV) and undergo PET scan within 12 weeks of SOC radiation therapy completion.

After completion of study intervention, patients are followed up every 8 weeks for 1 year followed by every 12 weeks for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥ 18 years of age.
* Patient must have a Karnofsky Performance Status ≥ 60%.
* Patient must have newly diagnosed GBM (must be IDH wild type), with pathologic proof, based on World Health Organization (WHO) 2021 criteria.
* Patient must be planning to receive standard-of-care treatment for newly diagnosed glioblastoma.
* Patient must have completed an MRI prior to the diagnostic surgery for GBM and have images available for upload into Transfer of Images and Data (TRIAD).
* Patient must have diagnostic surgery for GBM within 7 weeks prior to registration.
* Patient must have O6-Methylguanine-DNA Methyltransferase (MGMT) methylation status ordered at time of registration.
* Patient must have a post-operative (op) MRI completed within 3 weeks after diagnostic surgery for GBM and have images available for upload into TRIAD.
* Patient must have no contraindications to MRI, including injection of gadolinium-based contrast agents, and demonstrated ability to tolerate MRI on pre-surgical imaging.
* Patient must have no allergies to agents that may potentially be used for non-standard of care imaging (18F-fluciclovine, MR contrast).
* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the interventions being used.

  * All patients of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy.
  * A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From biomarker collection to death due to any cause, assessed up to 6 years
  Will use a two-sided log-rank test to compare the difference in OS between marker positive and marker negative participants using a significance level of 0.05.
Event free survival (EFS) | From biomarker collection until progression by Neurological Assessment in Neuro-Oncology (NANO) criteria or death, assessed up to 6 years
  NANO progression is defined as a ≥ 2 level worsening from baseline or best level of function in at least one domain or worsening to the highest score within ≥1 domain that is felt to be related to underlying tumor progression and not attributable to a comorbid event or change in concurrent medication. Will be based on the conditional power of a two-sided log-rank test for EFS between marker positive and marker negative participants using a significance level of 0.05.

SECONDARY OUTCOMES:
True disease progression and pseudo-progression (PsP) | Within 12 weeks post radiation therapy (XRT)
  The T3 MRI will be used to determine whether progressive enhancement seen within 12 weeks post-XRT was true progression or PsP.
Progression-free survival (PFS) | From surgery to the earlier of progression or death due to any cause, assessed up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel P Barboriak, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin, United States